CLINICAL TRIAL: NCT03756142
Title: Biomechanical Characterization of the Locomotion in Multiple Sclerosis Patients : Determination of Indicators of the Premature Degradation of the Orthostatic Posture, Gait Initiation and Walking
Brief Title: Biomechanical Characterization of the Locomotion in Multiple Sclerosis Patients
Acronym: WALKING-SEP
Status: Completed | Type: Observational
Sponsor: Lille Catholic University (Other)
Collaborators: Laboratoire d'Automatique, de Mécanique et d'Informatique Industrielles et Humaines (Unknown)
Responsible Party: Sponsor
Other Study IDs: RC-P0067
Record Dates: First submitted 2018-11-26; First posted 2018-11-28 (Actual); Last update posted 2024-03-06 (Actual); Status verified 2024-03

CONDITIONS: Multiple Sclerosis
Keywords: 3D analysis; Biomarkers; Rehabilition; Locomotion
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Multiple sclerosis patients: Analysis of orthostatic posture, initiation of walking and walking in MS patients with an EDSS between 0 and 4 (included) by a motion analysis system
  Interventions: Diagnostic Test: Motion Analysis
- Healthy volunteers: Analysis of orthostatic posture, initiation of walking and walking in a group of healthy volunteers
  Interventions: Diagnostic Test: Motion Analysis

INTERVENTIONS:
Diagnostic Test: Motion Analysis — Analysis of orthostatic posture, initiation of walking and walking by a motion analysis system

SUMMARY:
Multiple sclerosis (MS) is an inflammatory chronic disease of the central nervous system. Patients are suffering from balance and gait impairments at the early stage of the disease.

85 % of the MS patients report gait disorders, which impact their autonomy and their quality of life and increase the risk of fall.

The three-dimensional analysis of the walking by a motion capture system associated with force platforms allows the quantification of the complex walking disorders, to look for the cause, as well as side effects such as compensation strategies.

According to the 2006 report of the French National Authority for Health, the 3D analysis of walking is essential in chronic pathologies to evaluate and quantify gait disorders. This analysis allows the functional follow-up of the patients throughout their rehabilitation. Some studies, on a small and heterogeneous population of MS patients, showed changes during the walking concerning spatiotemporal, kinematic, dynamic parameters and muscular activation of lower limbs at early stages of the disease. Only two studies evaluate the joint power during walking in MS patients. However, these studies have some limits.

The 3D analysis of the walking proposed in this study would allow the biomechanical characterization of the gait impairments of MS patients through tasks such as walking, gait initiation and orthostatic posture. This methodology would contribute to adapt treatments and the rehabilitation care, at an early stage of the disease.

From a functional point of view, the gait initiation is an interesting dynamic task to be evaluated. Indeed, it represents the transition between the upright posture and the stabilized walking. Throughout this complex task, a stereotypical motor program is set up during a first phase of anticipatory postural adjustments, which allows the creation of dynamic conditions essential for the execution of the first step. The gait initiation is little documented for MS patients despite the risk of fall clinically highlighted. The articular power during the gait initiation was never estimated in MS patients. On the other hand, there is no study establishing correlations between the Expanded Disability Status Scale functional features and the impairments of the gait initiation.

ELIGIBILITY:
Inclusion Criteria for MS patients :

* EDSS < 4.5
* Stable disease for at least 6 weeks
* No injection of botulinum toxin in the past 4 months

no specific inclusion criteria for healthy volunteers

Exclusion Criteria for MS patients :

* Neurological disease other than MS
* Disabling pathologies of the locomotor apparatus
* Non-stabilized Respiratory, Cardiovascular disease
* Pregnant or breastfeeding women
* Patient with cognitive impairment
* Recent modification of MS treatment (<3 months)

Exclusion Criteria for Healthy Volunteers :

* Neurological disease
* Rheumatological disease
* Sprain of the lower limbs in the last 3 months
* Fracture of the lower limbs in the last year
* Pregnant or breastfeeding women

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with an early-stage of MS (cases) versus healthy controls who do not have MS.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2018-11-19 (Actual); Primary Completion 2020-01-07 (Actual); Study Completion 2020-01-07 (Actual)

PRIMARY OUTCOMES:
Kinematics of lower limbs articulations | at inclusion
  Kinematics of lower limbs will be performed by a motion analysis system. The analysis will be carried out with 4 infrared cameras, 2 force platforms, an electromyographic recording system, a computer system for signal analysis and data management. The optoelectronic system used is the 3D Vicon® system, which is based on passive stereovision. motive tasks (orthostatic posture, walking initiation, and the walking).

CONTACTS AND LOCATIONS:
Overall Officials: Caroline Massot, MD, Principal Investigator — GHICL
Locations (1):
- Hôpital Saint-Philibert, Lomme, France

IPD SHARING:
Plan to Share IPD: No